CLINICAL TRIAL: NCT07223905
Title: Motor-Cognitive Training for Motoric Cognitive Risk Syndrome
Acronym: VRTT for MCR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00161860
Record Dates: First submitted 2025-10-28; First posted 2025-11-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Motoric Cognitive Risk Syndrome

STUDY DESIGN:
Intervention Model Description: single-blind randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Treadmill Training (Experimental): The virtual reality treadmill training (VRTT) group will complete 18 training sessions over six weeks (three 1-hour sessions per week). Participants will perform prescribed tasks designed to challenge motor, cognitive, and motor-cognitive functions within a VR environment projected onto a screen in front of the treadmill (Fig 1). The VRTT system includes a conventional treadmill with a harness suspension system, camera-based motion capture (Intel RealSense, Santa Clara, CA), and a computer-generated simulation (GaitBetter, Tel Aviv, Israel). The camera tracks the participant's feet movements, which are displayed within the VR environment, allowing participants to see their feet navigating obstacles, pathways, and narrow corridors. Each session will include three walking bouts interspersed with rest breaks, targeting at least 40 minutes of active motor-cognitive training.
  Interventions: Behavioral: Virtual Reality Treadmill Training
- Treadmill Training (Active Comparator): Participants in the treadmill training (TT) intervention will follow a traditional TT program without feedback from the VR system. 70 The focus will be on increasing gait speed and distance, with no motor-cognitive training such as obstacle crossing or cognitive tasks while walking.
  Interventions: Behavioral: Treadmill Training

INTERVENTIONS:
Behavioral: Virtual Reality Treadmill Training — The Virtual Reality Treadmill Training (VRTT) group will complete 18 training sessions over six weeks (three 1-hour sessions per week). Participants will perform prescribed tasks designed to challenge motor, cognitive, and motor-cognitive functions within a VR environment projected onto a screen in front of the treadmill (Fig 1). The VRTT system includes a conventional treadmill with a harness suspension system, camera-based motion capture (Intel RealSense, Santa Clara, CA), and a computer-generated simulation (GaitBetter, Tel Aviv, Israel). The camera tracks the participant's feet movements, which are displayed within the VR environment, allowing participants to see their feet navigating obstacles, pathways, and narrow corridors. Each session will include three walking bouts interspersed with rest breaks, targeting at least 40 minutes of active motor-cognitive training.
  Arms: Virtual Reality Treadmill Training
Behavioral: Treadmill Training — Participants in the Treadmill Training (TT) intervention will follow a traditional TT program without feedback from the VR system. 70 The focus will be on increasing gait speed and distance, with no motor-cognitive training such as obstacle crossing or cognitive tasks while walking.
  Arms: Treadmill Training

SUMMARY:
The goal of this clinical trial is to investigate if combined motor-cognitive training can improve motor and cognitive symptoms in older adults with motoric cognitive risk syndrome. The main questions it aims to answer are:

* Does motor-cognitive training using a virtual reality treadmill improve gait speed?
* Does motor-cognitive training using a virtual reality treadmill improve cognitive functions?

Researchers will compare virtual reality treadmill training with treadmill training to see if virtual reality treadmill training works to improve motor and cognitive functions in older adults at risk of dementia

Participants will

* Complete 18 sessions (1 hour, 3x/week, 6 weeks) of either virtual reality treadmill training or treadmill training
* Complete a pre- and post-training assessment
* Wear an activity sensor for seven days prior to the pre-training assessment and for seven days after the post-training assessment.

DETAILED DESCRIPTION:
The objective of this single-blind randomized controlled trial is to compare the effects of combined motor-cognitive training using a virtual reality treadmill with motor training using a conventional treadmill in older adults with Motoric Cognitive Risk (MCR) syndrome. MCR is a geriatric condition characterized by slow gait speed and subjective cognitive complaints. The coexistence of motor and cognitive impairments in individuals with MCR significantly increases their risk of developing dementia. To date, randomized controlled trials investigating active interventions that simultaneously target both motor and cognitive functions remain scarce. This study will examine whether 18 training sessions, delivered over six weeks at a frequency of three 1-hour sessions per week, using a virtual reality treadmill lead to greater improvements in motor and cognitive outcomes compared to conventional treadmill training.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* English speaking
* Normal cognition (CDR=0)
* Meet MCR criteria
* Voluntary consent

Exclusion Criteria:

* Major chronic unstable disease or neurological condition (e.g., seizures)
* Diagnosed dementia
* Active psychiatric conditions
* Musculoskeletal conditions that affect walking for more than 2 minutes
* Severe visual or hearing impairments
* Sedating drugs (new use of narcotics or anxiolytics within the past month or chronic use that causes sedation)
* Currently engaged in other non-pharmacological interventions to improve cognition or walking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dual-task gait speed | From enrollment to the end of treatment at 6 weeks
  2 trials of 2-minute walking on a 10-meter walkway while completing auditory oddball task
Cognition | From enrollment to the end of treatment at 6 weeks
  Uniform Data Set (UDS) 4.0 global cognition composite score
Gait speed | From enrollment to the end of treatment at 6 weeks
  Gait speed on 4-meter walk test (4MWT)
Cognitive complaints | From enrollment to the end of treatment at 6 weeks
  Self-report of cognitive complaints based on memory item of the Geriatric Depression Scale (GDS): yes - no

SECONDARY OUTCOMES:
Dual task cost | From enrollment to the end of treatment at 6 weeks
  Motor and cognitive dual task cost defined using ((dual task - single task) / single task) * 100
Spatiotemporal gait characteristics | From enrollment to the end of treatment at 6 weeks
  Inertial Motion Units will collect spatiotemporal gait characteristics during single-task and dual-task walking
Cognitive domain scores | From enrollment to the end of treatment at 6 weeks
  Uniform Data Set 4.0 (UDS) cognitive domain scores
P3 event-related potential (ERP) | From enrollment to the end of treatment at 6 weeks
  P3 event-related potential (ERP) extracted from electroencephalography during oddball test
Mitochondrial function | From enrollment to the end of treatment at 6 weeks
  Mitochondrial functional index collected from blood serum

OTHER OUTCOMES:
Real-world physical activity and gait data | From enrollment to the end of treatment at 6 weeks
  Physical activity and gait data collected from activity sensors
Depression | From enrollment to the end of treatment at 6 weeks
  Scores on the Geriatric Depression Scale (GDS): range 0 - 15; higher score is worse
Health-related Quality of life | From enrollment to the end of treatment at 6 weeks
  Scores on Short Form 36 (SF-36): range 0 - 100; higher score is better
Frailty | From enrollment to the end of treatment at 6 weeks
  Scores on the Evaluative Frailty Index for Physical Activity (EFIPA): range 0 - 1; higher score is worse
Falls | From enrollment to the end of treatment at 6 weeks
  Self-report of falls via falls diaries
Resilience | From enrollment to the end of treatment at 6 weeks
  Brief Resilience Scale (BRS): range 6 - 30; higher scores are better

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No